CLINICAL TRIAL: NCT00516971
Title: The Use of Proton Pump Inhibitor for the Treatment of Non-erosive Gastro-oesophageal Reflux Disease in Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC1925-02; HARECCTR0500031
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Gastroesophageal Reflux
Keywords: Non-erosive reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole 20mg once daily

SUMMARY:
The purpose of this study is to evaluate the efficacy of proton pump inhibitor for the treatment of non-erosive reflux disease (NERD) in Chinese population. Studies from the western population have estimated a worldwide prevalence of gastro-oesophageal reflux disease from 10 to 20 %. Monthly symptoms of heartburn or acid regurgitation were found in 9.3% of subjects according to a population survey in Hong Kong. Most of these patients did not show evidence of erosive change during upper endoscopy. However, patients with NERD suffer from similar impairment of quality of life as patients with erosive oesophagitis and their symptoms are as severe as patients with erosive disease. Data on the use of proton pump inhibitor for the treatment of NERD in Chinese patients are scanty. Thus we want to perform a double-blind randomised placebo-controlled study to evaluate the efficacy of proton pump inhibitor for the treatment of NERD in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with age between 18 -80 years old,
* Patients with predominant symptoms of heartburn or acid regurgitation at least once weekly with no evidence of endoscopic pathology.

Exclusion Criteria:

* Patients under 18 or over 80 years of age,
* Symptoms of gastrointestinal bleeding,
* Patients who had previous upper gastrointestinal surgery,
* Patients with concomitant serious medical diseases,
* Patients who had received H2-receptor antagonists or proton pump inhibitors in the past 4 weeks,
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms assessment, quality of life. | 12 Weeks

SECONDARY OUTCOMES:
Compliance | 8 Weeks
Adverse effects | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ting Kin Cheung, Dr, Principal Investigator — Department of Medicine, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China